CLINICAL TRIAL: NCT00141765
Title: Myeloablative Chemotherapy With Stem Cell Rescue for Rare Poor-Prognosis Cancers
Brief Title: Study of High-Dose Chemotherapy With Bone Marrow or Stem Cell Transplant for Rare Poor-Prognosis Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, John Levine, MD, Professor of Pediatrics and of Internal Medicine, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9626; IRB 1996-195
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-05

CONDITIONS: Wilms Tumor; Fibrosarcoma; Carcinoma, Round Cell; Nasopharyngeal Cancer; Brain Tumor, Recurrent
MeSH Terms: conditions — Wilms Tumor; Fibrosarcoma; Carcinoma; Nasopharyngeal Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myeloablative Chemotherapy with Stem Cell Rescue (Experimental): Myeloablative Chemotherapy, followed by stem cell rescue
  Interventions: Procedure: Myeloablative Chemotherapy; Procedure: Stem Cell Rescue

INTERVENTIONS:
Procedure: Myeloablative Chemotherapy — High dose chemotherapy (carboplatin and thiotepa) transplant rescue
Procedure: Stem Cell Rescue — autologous stem cell transplantation

SUMMARY:
The purpose of this study is to determine whether very high dosages of chemotherapy will improve the chance of surviving cancer.

DETAILED DESCRIPTION:
This is a phase II trial designed to provide a transplant option for patients with rare poor-prognosis cancers. The protocol is only open to patients with metastatic or relapsed cancers for whom the probability of remaining free of progressive disease for one year after being brought into remission is < 25%. Patients eligible for this study have been diagnosed with a form of cancer that leads to death more than 75% of the time when treated with standard therapy doses of chemotherapy and/ or radiation therapy. Under this treatment intensification protocol the expectation is that the one year progression-free survival for this group of patients will rise to 40%. Patients eligible for this protocol will be followed for one year post-transplant. Patients alive and free of progressive disease at the end of this period will be considered successes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ineligible for other IRB-approved myeloablative regimens, be 21 years old or younger, and must have a histologically-confirmed Wilms' tumor, liver cancer, recurrent brain tumor of childhood, nasopharyngeal carcinoma, fibrosarcoma, desmoplastic small round cell tumor, germ cell tumor or other small round cell tumor, which:

  1. is metastatic and has < 25% cure rate with conventional treatment; or
  2. progressed after prior chemotherapy and has < 25% salvage rate with non-myeloablative therapies.
* Disease status: Within 3 weeks of initiation of this protocol, patients must:

  1. be in a complete or good partial remission (section 7.4); or
  2. have a "chemosensitive" tumor, which is defined as a > 50% decrease in at least one measurable tumor parameter attributable to prior chemotherapy, without evidence of progressive disease by any other parameter.
* Prior chemotherapy: Before entry to this protocol, patients must have derived maximal benefit from conventional, i.e., nonmyeloablative, doses of combination chemotherapy. Conventional therapy should be continued until either a complete remission is achieved, no further benefit from non-myeloablative dosing can be appreciated, or toxicity from conventional therapy is perceived as limiting in the absence of stem cell rescue. The cancer must be proven to be sensitive to alkylating agents. This means that, in addition to, or as part of, the appropriate chemotherapy protocol for the specific cancer in question, all patients must have received and responded to a minimum of:

  1. 2 courses of high-dose cyclophosphamide, totaling > 4200 mg/m2; or
  2. courses of high-dose ifosfamide totaling > 12 gm/m2.
  3. 1 course of "a)" above, plus 1 course of 'b)" above.
  4. Equivalent high dose alkylating agents as described in 3.3 a, b, and c.
* Patients must have adequate renal hepatic, and cardiac function (sections 4.4-4.6).
* Patients must meet at least one of the following stem cell requirements (Peripheral blood collection is to be preferred when available as an option):

  1. Harvested bone marrow must contain 1 x 108 nucleated cells per kg of body weight, or,
  2. Peripheral blood collection should include at least 2 x 106 CD34+ cells/kg.
* Informed consent must be signed indicating patient and/or parental awareness of the investigational nature of this program

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 1997-01; Primary Completion 2008-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Levine, MS MD, Principal Investigator — The Univeristy of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Myeloablative Chemotherapy With Stem Cell Rescue
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Myeloablative Chemotherapy With Stem Cell Rescue
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 6 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Progression Free Survival at 1 Year
Description: The primary outcome measure for this study was to improve the long-term disease-free survival of patients with rare cancers at high risk for lethal relapse.
Time Frame: 1 year post transplant
Measure: Number; unit: percentage of participants
Arm/Group | Myeloablative Chemotherapy With Stem Cell Rescue
Number analyzed (Participants) | 25
percentage of participants | 58

ADVERSE EVENTS:
Arm/Group | Myeloablative Chemotherapy With Stem Cell Rescue
Serious Adverse Events (participants affected / at risk) | 19/25
Other Adverse Events (participants affected / at risk) | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Myeloablative Chemotherapy With Stem Cell Rescue (N=25)
Mucocitis (Gastrointestinal disorders) | 10
Infection (Infections and infestations) | 11
Thrombocytopenia (Investigations) | 1
Death (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 6
Diarrhea (Gastrointestinal disorders) | 2
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2
Febrile Transfusion Reaction (Immune system disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Neutropenic Fever (Blood and lymphatic system disorders) | 2
Graft Failure (General disorders) | 1
Hypertension (Cardiac disorders) | 1
Disease Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure (Renal and urinary disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypcalcemia (Metabolism and nutrition disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Myeloablative Chemotherapy With Stem Cell Rescue (N=25)
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 5
Total Bilirubin (Investigations) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
ALK (Investigations) | 3
AST (Investigations) | 6
ALT (Investigations) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3
Esophagitis (Gastrointestinal disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Mucocitis (Gastrointestinal disorders) | 2
Hearing Loss (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes